CLINICAL TRIAL: NCT02865538
Title: Evaluation of the Pharmacokinetics and Safety of NT-814 in Post-Menopausal Women With Vasomotor Symptoms
Brief Title: Evaluation of the Pharmacokinetics and Safety of BAY3427080 (NT-814) in Post-Menopausal Women With Vasomotor Symptoms
Acronym: RELENT-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Nerre Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21681
Record Dates: First submitted 2016-08-03; First posted 2016-08-12 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Post-menopausal Vasomotor Symptoms
Keywords: Hot flashes; Post-menopausal
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BAY3427080 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (for BAY3427080)
- 50mg BAY3427080 (Experimental)
  Interventions: Drug: BAY3427080
- 100mg BAY3427080 (Experimental)
  Interventions: Drug: BAY3427080
- 150mg BAY3427080 (Experimental)
  Interventions: Drug: BAY3427080
- 300mg BAY3427080 (Experimental)
  Interventions: Drug: BAY3427080

INTERVENTIONS:
Drug: BAY3427080
  Other Names: NT-814
  Arms: 100mg BAY3427080; 150mg BAY3427080; 300mg BAY3427080; 50mg BAY3427080
Drug: Placebo (for BAY3427080)
  Arms: BAY3427080 Placebo

SUMMARY:
This is a multi-center, double-blind, randomized, placebo-controlled multiple ascending dose study in post-menopausal women with vasomotor symptoms. Single ascending doses of NT-814 will be investigated in 4 cohorts. Each cohort will comprise of 20 subjects. Subjects will be dosed for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female subjects experiencing frequent moderate to severe hot flashes.Menopause will be defined as:

  * 12 months of spontaneous amenorrhea;
  * OR at least 6 weeks' post-surgical bilateral oophorectomy with or without hysterectomy.

Exclusion Criteria:

* BMI > 35kg/m2.
* Any active comorbid disease, ECG or laboratory result deemed by the investigator to be clinically significant and which could impact safety during study conduct or that could interfere with the study evaluation, procedures or completion.
* Use of prohibited medications defined in the protocol.
* Inability or unwillingness to comply with study procedures or requirements.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Avail Clinical Research, DeLand, Florida
  - QPS/MRA (Miami Clinical Research), Miami, Florida
  - ICON Clinical Research Unit, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Trower M, Anderson RA, Ballantyne E, Joffe H, Kerr M, Pawsey S. Effects of NT-814, a dual neurokinin 1 and 3 receptor antagonist, on vasomotor symptoms in postmenopausal women: a placebo-controlled, randomized trial. Menopause. 2020 May;27(5):498-505. doi: 10.1097/GME.0000000000001500. PMID 32068688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 01 August 2016 (first subject, screening visit) and 28 March 2017 (last subject, last visit).
Pre-assignment Details: Overall 316 subjects were screened, of them 240 were screening failure. 76 subjects were randomized and assigned to treatment. 18 subjects were randomized to placebo and 58 subjects to BAY3427080 (NT-814) arms. 2 subjects discontinued the study .
Groups:
- Placebo Comparator: Placebo to match BAY3427080 capsules administered orally, daily, for 14 days. Number of placebo capsules to match active dose.
- 50 mg BAY3427080: 50mg of BAY3427080 to be administered as oral capsules, daily, for 14 days.
- 100 mg BAY3427080: 100 mg of BAY3427080 to be administered as oral capsules, daily, for 14 days
- 150 mg BAY3427080: 150 mg of BAY3427080 to be administered as oral capsules, daily, for 14 days.
- 300 mg of BAY3427080: 300 mg of BAY3427080 to be administered as oral capsules, daily, for 14 days.
Period: Overall Study
Arm/Group | Placebo Comparator | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg of BAY3427080
Started (76) | 18 | 15 | 15 | 15 | 13
Completed (74) | 17 | 15 | 14 | 15 | 13
Not Completed | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg of BAY3427080 | Total
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (4.08) | 55.9 (5.57) | 55.3 (5.43) | 56.7 (4.37) | 53.8 (3.88) | 55.4 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 15 | 15 | 13 | 76
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 8 | 10 | 9 | 50
  Not Hispanic or Latino | 5 | 5 | 7 | 5 | 4 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 4 | 2 | 2 | 14
  White | 16 | 11 | 11 | 13 | 11 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 73.25 (10.11) | 70.85 (11.82) | 73.47 (14.93) | 72.10 (7.10) | 72.73 (12.05) | 72.48 (11.20)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of BAY3427080
Description: Cmax is the maximum observed plasma concentration of BAY3427080 was presented. Blood samples were taken within 30 minutes prior to dose administration.
Time Frame: On Day 1, Day 7 (Pre-dose; 0.5; 1.0; 1.5; 2.0; 2.5; 3.0; 4.0; 5.0; 6.0; 8.0; 12.0; 24.0 hours) and on Day 14 (Pre-dose; 0.5; 1.0; 1.5; 2.0; 2.5; 3.0; 4.0; 5.0; 6.0; 8.0; 12.0; 24.0, 48.0, 72.0 hours)
Population: Participants who received placebo were not included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Placebo: Placebo to match BAY3427080 capsules administered orally, daily, for 14 days. Number of placebo capsules to match active dose.
- 300 mg BAY3427080: 300 mg BAY3427080 to be administered as oral capsules, daily, for 14 days.
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 0 | 15 | 15 | 15 | 13
ng/mL
  Day 1 |  | 502.62 (90.19) | 731.69 (110.58) | 911.48 (148.28) | 1576.01 (90.70)
  Day 7: number analyzed (Participants) | 0 | 14 | 15 | 15 | 13
  Day 7 |  | 548.60 (57.47) | 809.48 (116.58) | 1173.50 (95.14) | 2045.61 (152.87)
  Day 14: number analyzed (Participants) | 0 | 15 | 14 | 15 | 13
  Day 14 |  | 522.36 (87.88) | 841.42 (107.16) | 1188.19 (131.20) | 2851.83 (116.53)

2. Primary Outcome: Time to Reach Maximum Observed Drug Concentration in Plasma (Tmax) of BAY3427080
Description: Time of occurrence of Cmax.Time to reach maximum plasma concentration of BAY3427080 was presented. Blood samples for Tmax were taken within 30 minutes prior to dose administration.
Time Frame: as for outcome 1
Population: Participants who received placebo were not included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 0 | 15 | 15 | 15 | 13
hr
  Day 1 |  | 1.360 (40.01) | 1.320 (38.79) | 1.521 (41.95) | 1.471 (63.05)
  Day 7: number analyzed (Participants) | 0 | 14 | 15 | 15 | 13
  Day 7 |  | 1.432 (39.25) | 1.623 (43.19) | 1.536 (40.08) | 1.754 (56.18)
  Day 14: number analyzed (Participants) | 0 | 15 | 14 | 15 | 13
  Day 14 |  | 1.265 (46.32) | 1.445 (56.71) | 1.296 (23.35) | 1.342 (33.46)

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of BAY3427080
Description: AUC from time zero extrapolated to infinity of BAY3427080 was presented. AUC0-∞ was only estimated following the Day 1 dose.
Time Frame: Day 1 (pre-dose and post-dose (0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 5.0, 6.0, 8.0, 12.0 and 24.0 hours)
Population: Participants in PK population with available data are reported. Participants who received placebo were not included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 0 | 7 | 2 | 3 | 5
hr*ng/mL |  | 2018.68 (38.43) | 1545.58 (3.49) | 1151.87 (66.73) | 6249.52 (101.01)

4. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-τ) of BAY3427080
Description: Area under the concentration-time curve (AUC) from time zero to the time of the last quantifiable concentration of BAY3427080 was presented. Blood samples for (AUC0-τ) were taken within 30 minutes prior to dose administration.
Time Frame: as for outcome 1
Population: Participants who received placebo were not included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 0 | 15 | 15 | 15 | 13
hr*ng/mL
  Day 1 |  | 1400.167 (67.87) | 2341.882 (71.19) | 3012.793 (97.74) | 6527.569 (70.50)
  Day 7: number analyzed (Participants) | 0 | 14 | 15 | 15 | 13
  Day 7 |  | 2506.97 (48.05) | 4472.76 (63.83) | 6202.894 (43.92) | 12859.660 (85.47)
  Day 14: number analyzed (Participants) | 0 | 15 | 14 | 15 | 13
  Day 14 |  | 2341.55 (64.73) | 3542.41 (86.34) | 5163.500 (88.71) | 14822.860 (99.68)

5. Primary Outcome: Terminal Elimination Half-life (t½) of BAY3427080
Description: Terminal elimination half-life of BAY3427080 was presented. Blood samples were taken within 30 minutes prior to dose administration.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 0 | 7 | 2 | 8 | 11
hr
  Day 1: number analyzed (Participants) | 0 | 7 | 2 | 3 | 5
  Day 1 |  | 2.409 (34.15) | 1.903 (11.98) | 3.965 (45.94) | 3.142 (18.92)
  Day 7: number analyzed (Participants) | 0 | 2 | 2 | 3 | 1
  Day 7 |  | 2.443 (9.33) | 3.303 (21.20) | 3.482 (22.57) | 2.271
  Day 14: number analyzed (Participants) | 0 | 7 | 1 | 8 | 11
  Day 14 |  | 2.698 (21.64) | 2.042 | 21.593 (24.58) | 20.427 (22.85)

6. Primary Outcome: Apparent Clearance (CL/F) of BAY3427080
Description: Apparent clearance of BAY3427080 was presented. Blood samples were taken within 30 minutes prior to dose administration.
Time Frame: as for outcome 1
Population: Participants who received placebo were not included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 0 | 15 | 15 | 15 | 13
L/hr
  Day 1: number analyzed (Participants) | 0 | 7 | 2 | 3 | 5
  Day 1 |  | 24.769 (38.43) | 64.700 (3.49) | 130.223 (66.73) | 48.004 (101.01)
  Day 7: number analyzed (Participants) | 0 | 14 | 15 | 15 | 13
  Day 7 |  | 19.944 (48.05) | 22.358 (63.83) | 24.182 (43.92) | 23.329 (85.47)
  Day 14: number analyzed (Participants) | 0 | 15 | 14 | 15 | 13
  Day 14 |  | 21.353 (64.73) | 28.229 (86.34) | 29.050 (88.71) | 20.239 (99.68)

7. Primary Outcome: Number of Participants With Clinically Significant Abnormalities Detected Upon Physical Examination.
Description: A physician or appropriately qualified delegate conducted a full physical examination. Clinically significance was decided by investigator. The findings are presented as abnormal (clinically significant).
Time Frame: At day 14
Measure: Number; unit: Participants
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Participants | 1 | 0 | 2 | 1 | 2

8. Primary Outcome: Number of Participants With Clinically Significant Abnormalities on the 12-lead ECGs
Description: Reported results are cardiovascular system-examination findings at day 14. Clinically significance was decided by investigator. The findings are presented as abnormal (clinically significant).
Time Frame: At day 14
Measure: Number; unit: Participants
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Participants | 0 | 0 | 1 | 0 | 0

9. Primary Outcome: Number of Participants With Arrhythmias as Assessed by Continuous Holter Monitoring.
Description: Holter monitors were supplied by iCardiac Technologies. Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14 and remained in place until 24-hour assessments were completed.
Time Frame: Baseline (day -1) and day 14
Measure: Number; unit: Participants
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Participants
  Average Hourly Daytime Heart Rate < 50 bpm (daytime defined as 7 am-10 pm)(Day-1) | 0 | 0 | 1 | 0 | 0
  Frequent Supraventricular Premature Beats (APBs) (>100/24hrs) (Day-1) | 2 | 1 | 3 | 0 | 0
  Frequent Ventricular Ectopic Beats (VEs) (> 200/24hrs) (Day-1) | 1 | 4 | 1 | 0 | 2
  Other arrhythmias (Day-1) | 17 | 13 | 15 | 15 | 12
  Second Degree AV Block - Type I (Day-1) | 1 | 0 | 0 | 0 | 0
  Sinus Bradycardia (HR < 40 bpm)(Day-1) | 0 | 0 | 1 | 0 | 0
  SupraVentricular Tachycardia (lasting > 10 beats) (Day-1) | 4 | 5 | 4 | 2 | 1
  At least three monomorphic beats in a row (Day 14) | 0 | 0 | 0 | 1 | 0
  Average Hourly Daytime Heart Rate < 50 bpm (daytime defined as 7 am-10 pm) (Day 14) | 0 | 0 | 0 | 0 | 1
  Frequent Supraventricular Premature Beats (APBs) (>100/24hrs) (Day 14) | 1 | 0 | 0 | 0 | 0
  Frequent Ventricular Ectopic Beats (VEs) (> 200/24hrs) (Day 14) | 1 | 4 | 0 | 0 | 1
  Other arrhythmias (Day 14) | 18 | 14 | 13 | 15 | 13
  Presence of NSVT (Non-Sustained Ventricular Tachycardia) episodes (Day 14) | 0 | 0 | 0 | 1 | 0
  Second Degree AV Block - Type I (Day 14) | 2 | 0 | 0 | 0 | 0
  Second Degree AV Block - Type II(Day 14) | 1 | 0 | 0 | 1 | 0
  Sinus Bradycardia (HR < 40 bpm) | 0 | 0 | 0 | 1 | 0
  SupraVentricular Tachycardia (lasting > 10 beats (Day 14) | 3 | 3 | 1 | 1 | 1

10. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Diastolic Blood Pressure (Standing)
Description: Diastolic Blood Pressure was measured just prior to dosing (approx. 30 mins) in standing position.
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mmHg
  Baseline | 80.11 (4.702) | 76.07 (5.257) | 77.67 (11.462) | 78.93 (6.147) | 77.92 (9.768)
  Day 14 Change from Baseline | 1.11 (9.579) | 2.53 (5.540) | -0.07 (12.137) | 0.93 (7.216) | 1.62 (9.097)

11. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Diastolic Blood Pressure (Sitting)
Description: Diastolic Blood Pressure was measured just prior to dosing (approx. 30 mins) in sitting position.
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mmHg
  Baseline | 77.72 (6.542) | 74.27 (6.239) | 77.20 (10.705) | 74.80 (6.774) | 74.15 (8.245)
  Day 14 Change from Baseline | 0.11 (9.292) | -0.53 (6.906) | -0.79 (9.736) | 2.73 (9.384) | 1.77 (6.366)

12. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Systolic Blood Pressure (Standing)
Description: Systolic Blood Pressure was measured just prior to dosing (approx. 30 mins) in standing position.
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mmHg
  Baseline | 117.83 (10.733) | 114.60 (8.675) | 121.33 (17.867) | 118.87 (11.513) | 114.77 (15.095)
  Day 14 Change from Baseline | 5.11 (11.483) | 3.80 (13.311) | -4.43 (18.744) | 0.33 (12.234) | 5.62 (16.536)

13. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Systolic Blood Pressure (Sitting)
Description: Systolic Blood Pressure was measured just prior to dosing (approx. 30 mins) in sitting position.
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mmHg
  Baseline | 116.39 (11.304) | 113.80 (9.405) | 119.07 (15.931) | 117.20 (10.638) | 114.15 (14.288)
  Day 14 Change from Baseline | 4.17 (11.868) | 0.20 (10.359) | -2.79 (16.470) | 2.47 (16.890) | 5.62 (12.672)

14. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Pulse Rate
Description: Pulse rate was measured just prior to dosing (approx. 30 mins).
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
beats/min
  Baseline | 69.89 (8.629) | 66.00 (6.358) | 69.20 (9.966) | 68.40 (4.611) | 72.62 (7.136)
  Day 14 Change from Baseline | 1.06 (8.271) | -2.00 (8.027) | 0.14 (7.263) | 0.27 (8.388) | -11.00 (9.618)

15. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Respiratory Rate
Description: Respiratory rate was measured just prior to dosing (approx. 30 mins).
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
breaths/min
  Baseline | 15.39 (1.378) | 15.47 (1.727) | 15.73 (1.624) | 15.60 (1.502) | 15.85 (1.573)
  Day 14 Change from Baseline | -0.11 (2.220) | -0.40 (2.197) | 0.07 (1.940) | -0.43 (2.065) | -1.33 (1.923)

16. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Oxygen Saturation
Description: Oxygen Saturation was measured just prior to dosing (approx. 30 mins).
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: Percentage of Oxygen satuartion
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Percentage of Oxygen satuartion
  Baseline | 98.50 (1.098) | 98.40 (1.404) | 97.87 (1.727) | 97.67 (1.496) | 97.31 (1.251)
  Day 14 Change from Baseline | -0.61 (1.539) | -0.73 (1.486) | 0.29 (2.091) | 0.20 (1.424) | 0.38 (1.193)

17. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Oral Body Temperature
Description: Temperature was measured just prior to dosing (approx. 30 mins).
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: Degree Celius
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Degree Celius
  Baseline | 36.77 (0.190) | 36.65 (0.155) | 36.79 (0.162) | 36.71 (0.168) | 36.77 (0.361)
  Day 14 Change from Baseline | -0.04 (0.243) | 0.06 (0.172) | -0.09 (0.264) | -0.01 (0.239) | -0.05 (0.458)

18. Primary Outcome: Change From Baseline at Day 14 in Vital Signs: Weight
Description: Weight was measured just prior to dosing (approx. 30 mins).
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Kilograms
  Baseline | 73.25 (10.115) | 70.85 (11.821) | 73.47 (14.934) | 72.10 (7.104) | 72.73 (12.047)
  Day 14 Change from Baseline | 0.36 (1.034) | 0.51 (0.983) | 0.24 (0.916) | 0.15 (0.926) | 0.01 (0.704)

19. Primary Outcome: Change From Baseline at Day 15 for Laboratory Hormones Results : Adrenocorticotropic Hormone (ADTH) and Estradiol.
Description: Blood samples for the assessment of ACTH and Estradiol were collected upon participants admission to the unit.
Time Frame: Baseline and day 15
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
pmol/L
  Baseline (ADTH) | 5.34 (3.402) | 4.17 (1.991) | 3.87 (2.361) | 3.55 (2.360) | 3.27 (2.011)
  Day 15 Change from Baseline (ADTH) | -0.49 (3.333) | -0.68 (2.035) | 0.84 (1.914) | 1.04 (3.059) | 1.67 (3.059)
  Baseline (Estradiol) | 57.33 (43.236) | 59.49 (40.129) | 35.02 (25.556) | 43.83 (31.270) | 62.42 (42.589)
  Day 15 Change from Baseline (Estradiol): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 15 Change from Baseline (Estradiol) | 22.43 (141.618) | 13.21 (80.704) | 0.53 (3.172) | 1.96 (12.394) | -9.02 (87.480)

20. Primary Outcome: Change From Baseline at Day 15 for Laboratory Hormones Results: Follicle Stimulating Hormone
Description: Blood samples for the assessment of Follicle Stimulating were collected upon participants admission to the unit.
Time Frame: Baseline and day 15
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
IU/L
  Baseline | 76.01 (23.122) | 100.87 (36.813) | 77.78 (20.132) | 88.77 (42.251) | 70.59 (17.046)
  Day 15 Change from Baseline | 5.98 (13.072) | -2.29 (20.948) | 4.09 (8.353) | 6.73 (6.904) | 8.92 (13.409)

21. Primary Outcome: Change From Baseline at Day 15 for Laboratory Hormones Results : Triiodothyronine Uptake
Description: Blood samples for the assessment of Triiodothyronine were collected upon participants admission to the unit.
Time Frame: Baseline and day 15
Population: Participants in PK analysis set with evaluable data for this outcome measure presented.
Measure: Mean (Standard Deviation); unit: Percentage of T Uptake
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 0
Percentage of T Uptake
  Baseline: number analyzed (Participants) | 5 | 4 | 8 | 7 | 0
  Baseline | 32.300 (3.5623) | 30.800 (2.4712) | 30.838 (1.7968) | 30.671 (1.3060) |
  Day 15 Change from Baseline | -0.720 (0.7662) | -0.700 (0.2944) | 0.143 (0.7115) | 0.443 (1.0130) |

22. Primary Outcome: Change From Baseline at Day 15 for Laboratory Hormones Results: Thyrotropin
Description: Blood samples for the assessment of Thyrotropin were collected upon participants admission to the unit.
Time Frame: Baseline and day 15
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mIU/L
  Baseline | 2.658 (1.7584) | 1.800 (0.9830) | 2.451 (1.4811) | 2.785 (1.1449) | 2.330 (1.2658)
  Day 15 Change from Baseline | -0.959 (1.3501) | -0.571 (0.8148) | -0.648 (0.5903) | -0.823 (1.0604) | -0.616 (1.1375)

23. Primary Outcome: Change From Baseline at Day 15 for Laboratory Hormones Results : Cortisol, Testosterone, Thyroxine and Triiodothyronine
Description: Blood samples for the assessment of Cortisol, Testosterone, Thyroxine and Triiodothyronine were collected upon participants admission to the unit.
Time Frame: Baseline and day 15
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
nmol/L
  Baseline (Cortisol) | 348.60 (156.496) | 337.16 (177.507) | 345.91 (173.302) | 251.66 (144.743) | 230.42 (74.560)
  Day 15 Change from Baseline (Cortisol): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 15 Change from Baseline (Cortisol) | 15.94 (193.564) | -23.32 (172.685) | 68.05 (170.121) | 92.02 (159.464) | 127.20 (208.452)
  Baseline (Testosterone) | 0.744 (0.3850) | 0.666 (0.6230) | 0.517 (0.2317) | 0.433 (0.2961) | 0.611 (0.4271)
  Day 15 Change from Baseline (Testosterone): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 15 Change from Baseline (Testosterone) | 0.057 (0.3567) | 0.024 (0.2578) | 0.696 (0.3367) | 0.480 (0.4589) | 0.524 (0.2905)
  Baseline(Thyroxine) | 95.44 (14.576) | 95.66 (15.203) | 96.11 (14.645) | 86.41 (16.116) | 94.16 (22.180)
  Day 15 Change from Baseline(Thyroxine) | -3.78 (14.771) | -1.28 (8.127) | -10.67 (26.324) | 6.53 (9.546) | 0.88 (13.720)
  Baseline(Triiodothyronine): number analyzed (Participants) | 12 | 11 | 7 | 8 | 7
  Baseline(Triiodothyronine) | 1.865 (0.14131) | 2.060 (0.3174) | 1.980 (0.2916) | 1.776 (0.4510) | 2.163 (0.6008)
  Day 15 Change from Baseline (Triiodothyronine): number analyzed (Participants) | 12 | 11 | 7 | 8 | 7
  Day 15 Change from Baseline (Triiodothyronine) | -0.190 (0.3171) | -0.141 (0.2742) | -0.407 (0.2180) | -0.148 (0.1883) | -0.416 (0.5359)

24. Primary Outcome: Change From Baseline at Day 14 for Clinical Laboratory Parameters LIPIDS : Cholesterol, Triglycerides, HDL Cholesterol and LDL Cholesterol.
Description: Blood samples for the assessment of Cholesterol, Triglycerides,high-density lipoprotein (HDL)Cholesterol and low-density lipoprotein (LDL) Cholesterol were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mmol/L
  Baseline (Cholesterol) | 5.434 (1.0223) | 5.471 (0.6592) | 5.391 (0.7346) | 5.804 (0.6462) | 5.393 (0.9008)
  Day 14 Change from Baseline (Cholesterol): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Cholesterol) | 0.088 (0.8629) | -0.061 (0.4761) | -0.205 (0.8981) | -0.185 (0.6386) | -0.321 (0.6790)
  Baseline (Triglycerides) | 1.163 (0.5796) | 1.185 (0.5036) | 1.131 (0.5889) | 1.329 (0.6245) | 1.353 (0.5540)
  Day 14 Change from Baseline (Triglycerides): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Triglycerides) | 0.048 (0.4936) | -0.071 (0.4725) | -0.116 (0.5247) | -0.029 (0.4178) | -0.172 (0.5633)
  Baseline(HDL Cholesterol) | 1.717 (0.4525) | 1.879 (0.4052) | 1.7444 (0.6563) | 1.768 (0.4716) | 1.449 (0.2752)
  Day 14 Change from Baseline( HDL Cholesterol): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline( HDL Cholesterol) | -0.167 (0.2824) | -0.219 (0.2015) | -0.056 (0.2559) | -0.147 (0.1546) | -0.158 (0.3132)
  Baseline( LDL Cholesterol) | 3.226 (1.0485) | 3.125 (0.8436) | 3.172 (0.7654) | 3.625 (0.7188) | 3.552 (1.1088)
  Day 14 Change from Baseline ( LDL Cholesterol): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline ( LDL Cholesterol) | -0.013 (0.3926) | 0.184 (0.2958) | -0.119 (0.6747) | -0.038 (0.6490) | -0.053 (0.5944)

25. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Immature Granulocytes.
Description: Blood samples for the assessment of Neutrophils/Leukocytes, Lymphocytes /Leukocytes, Monocytes/Leukocytes, Eosinophils/Leukocytes, Basophils/Leukocytes and Immature Granulocytes/ Leukocytes were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: Percentage of total white blood cells
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Percentage of total white blood cells
  Baseline (Neutrophils/ Leukocytes) | 56.53 (7.700) | 53.31 (4.994) | 55.65 (8.318) | 54.78 (8.610) | 50.92 (10.316)
  Day 14 Change from Baseline (Neutrophils/ Leukocytes): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Neutrophils/ Leukocytes) | -0.29 (7.788) | 2.41 (6.119) | -0.50 (5.047) | -0.98 (7.116) | -2.69 (10.614)
  Baseline (Lymphocytes/ Leukocytes) | 32.40 (7.098) | 35.57 (5.439) | 33.33 (8.024) | 34.33 (7.444) | 36.78 (10.446)
  Day 14 Change from Baseline(Lymphocytes / Leukocytes): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Lymphocytes / Leukocytes) | 0.18 (5.791) | -2.46 (5.667) | -0.11 (4.763) | 0.59 (5.835) | 2.75 (10.926)
  Baseline ( Monocytes / Leukocytes ) | 7.58 (1.592) | 7.47 (1.379) | 7.62 (1.591) | 7.71 (1.762) | 8.62 (3.276)
  Day 14 Change from Baseline( Monocytes/ Leukocytes): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline( Monocytes/ Leukocytes) | 0.22 (1.947) | -0.15 (1.751) | 0.65 (1.291) | 0.05 (2.758) | 0.22 (3.850)
  Baseline ( Eosinophils/ Leukocytes) | 2.83 (2.433) | 3.04 (3.352) | 2.64 (1.422) | 2.61 (1.170) | 3.05 (1.979)
  Day 14 Change from Baseline(Eosinophils/ Leukocytes): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Eosinophils/ Leukocytes) | 0.02 (1.316) | 0.29 (0.961) | 0.06 (0.794) | 0.33 (0.538) | -0.24 (1.189)
  Baseline(Basophils/ Leukocytes) | 0.61 (0.263) | 0.55 (0.177) | 0.66 (0.295) | 0.51 (0.223) | 0.56 (0.373)
  Day 14 Change from Baseline (Basophils/ Leukocytes): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Basophils/ Leukocytes) | -0.13 (0.181) | -0.07 (0.111) | -0.14 (0.122) | 0.01 (0.209) | -0.05 (0.307)
  Baseline( Immature Granulocytes/ Leukocytes): number analyzed (Participants) | 6 | 4 | 8 | 7 | 6
  Baseline( Immature Granulocytes/ Leukocytes) | 0.15 (0.084) | 0.25 (0.100) | 0.20 (0.151) | 0.13 (0.111) | 0.15 (0.084)
  Day 14 Change from Baseline( Immature Granulocytes/ Leukocytes): number analyzed (Participants) | 6 | 4 | 7 | 7 | 6
  Day 14 Change from Baseline( Immature Granulocytes/ Leukocytes) | 0.03 (0.082) | -0.05 (0.100) | 0.09 (0.157) | 0.00 (0.183) | 0.03 (0.137)

26. Primary Outcome: Change From Baseline at Day 14 for Clinical Laboratory Parameters HEMATOLOGY: Leukocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, Immature Granulocytes and Platelets.
Description: Blood samples for the assessment of Leukocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, Immature Granulocytes and Platelets were collected upon participant's admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: 10^9*cells/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
10^9*cells/L
  Baseline( Leukocytes) | 6.73 (1.372) | 6.54 (1.613) | 6.75 (1.245) | 6.78 (1.307) | 6.60 (1.896)
  Day 14 Change from Baseline( Leukocytes) | -0.60 (1.299) | -0.27 (1.134) | -0.34 (0.686) | -0.80 (1.011) | -0.06 (1.650)
  Baseline (Neutrophils) | 3.847 (1.0899) | 3.493 (0.9737) | 3.779 (0.9332) | 3.745 (0.9686) | 3.394 (1.3264)
  Day 14 Change from Baseline (Neutrophils ): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Neutrophils ) | -0.374 (1.1794) | 0.072 (0.7422) | -0.246 (0.5487) | -0.539 (0.9017) | -0.186 (1.4444)
  Baseline (Lymphocytes) | 2.148 (0.4905) | 2.341 (0.7009) | 2.242 (0.6199) | 2.320 (0.6467) | 2.429 (0.9032)
  Day 14 Change from Baseline (Lymphocytes): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Lymphocytes) | -0.172 (0.2900) | -0.301 (0.5336) | -0.107 (0.3652) | -0.237 (0.3901) | 0.142 (0.6749)
  Baseline ( Monocytes) | 0.499 (0.0984) | 0.479 (0.1051) | 0.505 (0.0990) | 0.524 (0.1410) | 0.534 (0.1552)
  Day 14 Change from Baseline( Monocytes) | -0.033 (0.1117) | -0.030 (0.1324) | 0.019 (0.0895) | -0.057 (0.1941) | 0.002 (0.1643)
  Baseline ( Eosinophils) | 0.202 (0.2325) | 0.185 (0.1814) | 0.177 (0.1090) | 0.177 (0.0954) | 0.208 (0.1592)
  Day 14 Change from Baseline(Eosinophils): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Eosinophils) | -0.017 (0.0995) | 0.021 (0.0719) | -0.006 (0.0549) | 0.005 (0.0436) | -0.028 (0.1155)
  Baseline(Basophils) | 0.041 (0.0305) | 0.031 (0.0264) | 0.028 (0.0321) | 0.027 (0.0301) | 0.030 (0.327)
  Day 14 Change from Baseline(Basophils): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Basophils) | -0.008 (0.0148) | -0.007 (0.0090) | -0.001 (0.0305) | -0.010 (0.0259) | -0.002 (0.0060)
  Baseline( Immature Granulocytes): number analyzed (Participants) | 6 | 4 | 8 | 7 | 6
  Baseline( Immature Granulocytes) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 14 Change from Baseline( Immature Granulocytes): number analyzed (Participants) | 6 | 4 | 7 | 7 | 6
  Day 14 Change from Baseline( Immature Granulocytes) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Baseline (Platelets ) | 263.4 (59.66) | 249.1 (61.67) | 269.8 (61.40) | 261.9 (46.91) | 258.2 (52.57)
  Day 14 Change from Baseline(Platelets ): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Platelets ) | 8.1 (17.77) | 4.5 (33.83) | 13.5 (29.67) | 21.6 (24.58) | 20.8 (74.35)

27. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Hemoglobin and Erythrocytes Mean Corpuscular Hemoglobin Concentration
Description: Blood samples for the assessment of Hemoglobin and Erythrocytes Mean Corpuscular Hemoglobin (HB)concentration were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
g/L
  Baseline (Hemoglobin) | 128.9 (8.53) | 132.4 (10.64) | 128.7 (7.82) | 127.7 (8.60) | 132.2 (12.60)
  Day 14 Change from Baseline (Hemoglobin): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Hemoglobin) | -11.8 (4.99) | -9.0 (7.14) | -14.6 (5.98) | -13.9 (4.66) | -12.1 (6.58)
  Baseline (Erythrocytes Mean Corpuscular HB concentration ): number analyzed (Participants) | 15 | 11 | 12 | 13 | 11
  Baseline (Erythrocytes Mean Corpuscular HB concentration ) | 328.5 (10.30) | 335.2 (9.42) | 329.0 (10.22) | 328.2 (7.51) | 326.8 (10.27)
  Day 14 Change from Baseline (Erythrocytes Mean Corpuscular HB concentration): number analyzed (Participants) | 15 | 11 | 11 | 13 | 11
  Day 14 Change from Baseline (Erythrocytes Mean Corpuscular HB concentration) | -0.4 (5.21) | -2.5 (2.34) | -2.3 (6.94) | -0.8 (3.41) | 3.2 (4.62)

28. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Erythrocytes
Description: Blood samples for the assessment of Erythrocytes were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: 10^12*cells/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
10^12*cells/L
  Baseline | 4.467 (0.2503) | 4.525 (0.2212) | 4.459 (0.2962) | 4.365 (0.3678) | 4.518 (0.2368)
  Day 14 Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline | -0.421 (0.1750) | -0.301 (0.2694) | -0.511 (0.2111) | -0.485 (0.1903) | -0.425 (0.2297)

29. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Erythrocytes Mean Corpuscular Volume and Mean Platelet Volume.
Description: Blood samples for the assessment of Erythrocytes Mean Corpuscular Volume and Mean Platelet Volume were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
fL
  Baseline (Erythrocytes Mean Corpuscular Volume ) | 87.87 (5.707) | 87.69 (3.890) | 87.71 (4.717) | 89.42 (6.744) | 88.63 (3.150)
  Day 14 Change from Baseline (Erythrocytes Mean Corpuscular Volume ): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Erythrocytes Mean Corpuscular Volume ) | 0.44 (1.155) | 0.11 (0.799) | 0.47 (0.967) | 0.49 (1,691) | -0.27 (0.659)
  Baseline (Mean Platelet Volume): number analyzed (Participants) | 15 | 11 | 12 | 13 | 11
  Baseline (Mean Platelet Volume) | 9.79 (0.809) | 9.91 (1.608) | 10.22 (1.565) | 10.19 (1.005) | 10.05 (1.179)
  Day 14 Change from Baseline (Mean Platelet Volume): number analyzed (Participants) | 15 | 11 | 11 | 13 | 11
  Day 14 Change from Baseline (Mean Platelet Volume) | -0.14 (0.448) | 0.08 (0.412) | -0.24 (0.220) | -0.37 (0.403) | -0.06 (0.216)

30. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples for the assessment of Erythrocytes Mean Corpuscular Hemoglobin were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
pg
  Baseline: number analyzed (Participants) | 15 | 11 | 12 | 13 | 11
  Baseline | 28.89 (2.517) | 29.50 (1.803) | 28.79 (2.217) | 29.39 (2.511) | 28.89 (1.759)
  Day 14 Change from Baseline: number analyzed (Participants) | 15 | 11 | 11 | 13 | 11
  Day 14 Change from Baseline | 0.09 (0.494) | -0.19 (0.263) | 0.03 (0.486) | 0.15 (0.532) | 0.17 (0.317)

31. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Erythrocytes Distribution Width.
Description: Blood samples for the assessment of Erythrocytes Distribution Width were collected upon participants admission to the unit. Erythrocytes distribution width (in percentage) = 1 SD of Erythrocyte volume/MCV x 100%
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: Percentage of Erythrocyte volume
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Percentage of Erythrocyte volume
  Baseline: number analyzed (Participants) | 15 | 11 | 12 | 13 | 11
  Baseline | 27.81 (15.478) | 25.52 (15.413) | 35.82 (16.476) | 30.59 (16.089) | 31.48 (17.013)
  Day 14 Change from Baseline: number analyzed (Participants) | 15 | 11 | 11 | 13 | 11
  Day 14 Change from Baseline | -0.15 (0.916) | 0.49 (0.863) | -0.05 (1.878) | -0.61 (0.696) | -0.68 (0.778)

32. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters HEMATOLOGY: Hematocrit.
Description: Blood samples for the assessment of Hematocrit were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: Volume percentage
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Volume percentage
  Baseline | 39.18 (1.976) | 39.63 (2.461) | 38.99 (1.788) | 38.85 (1.990) | 40.02 (2.646)
  Day 14 Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline | -3.51 (1.307) | -2.45 (2.106) | -4.20 (1.877) | -4.13 (1.431) | -3.86 (2.163)

33. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters CHEMISTRY: Protein and Albumin.
Description: Blood samples for the assessment of Protein and Albumin were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
g/L
  Baseline (Protein) | 71.8 (4.54) | 72.2 (4.13) | 74.3 (4.25) | 70.5 (4.84) | 69.2 (4.22)
  Day 14 Change from Baseline(Protein): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Protein) | -4.0 (3.11) | -2.5 (4.39) | -6.9 (4.89) | -4.1 (2.64) | -2.5 (3.10)
  Baseline(Albumin) | 42.9 (6.75) | 44.3 (1.84) | 44.4 (2.53) | 44.7 (2.53) | 43.2 (2.67)
  Day 14 Change from Baseline (Albumin): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Albumin) | -0.6 (6.42) | -2.5 (2.42) | -3.2 (2.08) | 0.3 (2.05) | -1.8 (2.44)

34. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters CHEMISTRY: Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Gamma Glutamyl Transferase and Creatine Kinase
Description: Blood samples for the assessment of Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Gamma Glutamyl Transferase and Creatine Kinase were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
ukat/L
  Baseline (Alkaline Phosphatase) | 1.587 (0.4829) | 1.397 (0.3233) | 1.364 (0.3219) | 1.397 (0.3271) | 1.407 (0.4417)
  Day 14 Change from Baseline (Alkaline Phosphatase): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Alkaline Phosphatase) | -0.129 (0.3411) | -0.130 (0.2054) | -0.172 (0.1533) | -0.203 (0.2576) | -0.131 (0.2958)
  Baseline(Alanine Aminotransferase) | 0.295 (0.1302) | 0.331 (0.1494) | 0.279 (0.1151) | 0.313 (0.1281) | 0.413 (0.1755)
  Day 14 Change from Baseline (Alanine Aminotransferase): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Alanine Aminotransferase) | 0.108 (0.4103) | -0.049 (0.1053) | 0.049 (0,2099) | -0.016 (0.1391) | 0.052 (0.3923)
  Baseline (Aspartate Aminotransferase) | 0.344 (0.0760) | 0.355 (0.0632) | 0.343 (0.0950) | 0.352 (0.0737) | 0.401 (0.1976)
  Day 14 Change from Baseline (Aspartate Aminotransferase): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Aspartate Aminotransferase) | 0.041 (0.2197) | -0.035 (0.0542) | -0.032 (0.1030) | -0.009 (0.0743) | -0.032 (0.2851)
  Baseline (Gamma Glutamyl Transferase) | 0.309 (0.1740) | 0.324 (0.2085) | 0.397 (0.2111) | 0.561 (0.7998) | 0.372 (0.2272)
  Day 14 Change from Baseline (Gamma Glutamyl Transferase): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Gamma Glutamyl Transferase) | 0.101 (0.3890) | -0.035 (0.0980) | 0.001 (0.1606) | -0.190 (0.4620) | 0.015 (0.1959)
  Baseline (Creatine Kinase) | 1.957 (0.8872) | 2.047 (1.0146) | 1.907 (1.1933) | 1.895 (1.2638) | 1.886 (1.1854)
  Day 14 Change from Baseline (Creatine Kinase): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Creatine Kinase) | 0.021 (0.9758) | -0.260 (0.4338) | -0.252 (0.5078) | -0.038 (0.5689) | -0.269 (0.5032)

35. Primary Outcome: Change From Baseline at Day 14 for Laboratory Parameters CHEMISTRY: Urate, Bilirubin and Creatinine.
Description: Blood samples for the assessment of Urate, Bilirubin and Creatinine were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
umol/L
  Baseline (Urate): number analyzed (Participants) | 6 | 4 | 8 | 7 | 6
  Baseline (Urate) | 297.43 (41.896) | 318.23 (20.323) | 261.74 (57.222) | 275.34 (75.528) | 212.17 (52.885)
  Day 14 Change from Baseline (Urate): number analyzed (Participants) | 6 | 4 | 7 | 7 | 6
  Day 14 Change from Baseline (Urate) | -11.90 (41.380) | -2.95 (28.511) | 2.57 (19.706) | -12.76 (28.636) | -7.93 (44.269)
  Baseline (Bilirubin) | 7.61 (3.500) | 8.44 (3.640) | 7.19 (2.932) | 6.96 (2.652) | 7.23 (3.305)
  Day 14 Change from Baseline(Bilirubin): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Bilirubin) | -1.25 (3.225) | -1.15 (2.654) | -1.00 (1.886) | -0.01 (2.599) | 0.40 (3.069)
  Baseline(Creatinine) | 71.162 (11.3215) | 67.125 (8.0711) | 65.121 (9.8867) | 67.891 (9.1636) | 11.844 (8.9096)
  Day 14 Change from Baseline(Creatinine): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline(Creatinine) | 2.652 (6.4810) | -1.885 (7.8090) | -4.168 (7.6761) | -1.297 (6.6136) | -3.605 (5.6665)

36. Primary Outcome: Change From Baseline at Day 14 for Clinical Laboratory Parameters CHEMISTRY: Sodium, Potassium, Chloride, Bicarbonate, Calcium, Phosphate, Glucose, Magnesium and Urea Nitrogen.
Description: Blood samples for the assessment of Sodium, Potassium, Chloride, Bicarbonate, Calcium, Phosphate, Glucose, Magnesium and Urea Nitrogen were collected upon participant's admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mmol/L
  Baseline (Sodium) | 140.7 (2.93) | 140.3 (2.05) | 140.0 (1.65) | 142.3 (3.01) | 140.0 (2.83)
  Day 14 Change from Baseline (Sodium): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Sodium) | -0.9 (2.91) | -0.7 (2.97) | -0.5 (2.28) | -2.5 (3.23) | 0.7 (3.47)
  Baseline (Potassium) | 4.41 (0.375) | 4.22 (0.246) | 4.29 (0.374) | 4.49 (0.380) | 4.14 (0.421)
  Day 14 Change from Baseline (Potassium): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Potassium) | 0.06 (0.478) | 0.22 (0.323) | 0.15 (0.427) | -0.06 (0.408) | 0.31 (0.614)
  Baseline (Chloride) | 102.8 (2.94) | 102.4 (3.79) | 100.7 (2.32) | 102.7 (2.84) | 101.4 (1.56)
  Day 14 Change from Baseline ( Chloride): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline ( Chloride) | -1.2 (3.20) | 0.4 (3.16) | 1.1 (1.69) | -1.1 (3.02) | 0.8 (2.88)
  Baseline (Bicarbonate) | 26.39 (2.615) | 26.60 (2.131) | 27.47 (1.642) | 26.20 (1.699) | 27.62 (3.641)
  Day 14 Change from Baseline (Bicarbonate): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Bicarbonate) | 1.11 (3.660) | -0.93 (3.575) | 1.00 (3.088) | 2.00 (2.204) | 0.31 (2.626)
  Baseline (Calcium) | 2.421 (0.0803) | 2.401 (0.0730) | 2.515 (0.0998) | 2.411 (0.0622) | 2.382 (0.0928)
  Day 14 Change from Baseline (Calcium): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Calcium) | -0.032 (0.1198) | -0.044 (0.1355) | -0.144 (0.1147) | -0.049 (0.0630) | -0.052 (0.1103)
  Baseline (Phosphate) | 1.240 (0.1510) | 1.249 (0.1277) | 1.268 (0.1269) | 1.280 (0.1115) | 1.272 (0.1544)
  Day 14 Change from Baseline (Phosphate): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Phosphate) | 0.026 (0.1602) | -0.045 (0.1457) | -0.052 (0.1096) | 0.027 (0.1389) | -0.038 (0.2171)
  Baseline (Glucose) | 5.457 (0.6417) | 5.521 (0.4157) | 5.349 (0.4957) | 5.483 (0.3943) | 5.456 (0.4401)
  Day 14 Change from Baseline (Glucose): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Glucose) | -0.113 (0.9083) | -0.278 (0.4006) | -0.173 (0.3412) | -0.098 (0.4245) | 0.025 (0.3063)
  Baseline (Magnesium) | 0.893 (0.0732) | 0.885 (0.0588) | 0.881 (0.0675) | 0.905 (0.0703) | 0.896 (0.0836)
  Day 14 Change from Baseline (Magnesium): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Magnesium) | -0.009 (0.0460) | 0.001 (0.0387) | 0.001 (0.0529) | 0.006 (0.0484) | -0.027 (0.0696)
  Baseline (Urea Nitrogen) | 5.59 (1.230) | 5.47 (1.337) | 4.67 (1.274) | 5.30 (1.198) | 5.21 (1.393)
  Day 14 Change from Baseline (Urea Nitrogen): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Urea Nitrogen) | 0.14 (2.359) | -0.14 (1.070) | 0.20 (0.826) | 0.00 (1.442) | -0.38 (1.488)

37. Primary Outcome: Laboratory Parameters CHEMISTRY: Glomerular Filtration Rate African at Baseline
Description: Blood samples for the assessment of Glomerular Filtration Rate African were collected upon participants admission to the unit.
Time Frame: At Baseline
Population: Participants with available data reported. Baseline is the last available measurement prior to the first dose of study drug.
Measure: Mean (Standard Deviation); unit: mL/sec/1.73m^2
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mL/sec/1.73m^2 | 1.628 (0.2347) | 1.759 (0.1592) | 1.580 (0.1846) | 1.557 (0.1553) | 1.666 (0.1885)

38. Primary Outcome: Laboratory Parameters CHEMISTRY: Glomerular Filtration Rate Caucasian at Baseline
Description: Blood samples for the assessment of Glomerular Filtration Rate Caucasian were collected upon participants admission to the unit.
Time Frame: At Baseline
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mL/sec/1.73m^2
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
mL/sec/1.73m^2 | 1.343 (0.1955) | 1.450 (0.1265) | 1.300 (0.1503) | 1.290 (0.1273) | 1.378 (0.1482)

39. Primary Outcome: Change From Baseline at Day 14 for COAGULATION: Prothrombin International Normalized Ratio (INR)
Description: Blood samples for the assessment of Prothrombin International Normalized Ratio were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: INR
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
INR
  Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Baseline | 0.993 (0.0428) | 1.013 (0.0552) | 1.007 (0.0482) | 0.991 (0.0465) | 0.993 (0.0645)
  Day 14 Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline | -0.007 (0.0546) | -0.038 (0.0471) | 0.016 (0.0665) | 0.013 (0.0359) | 0.057 (0.2311)

40. Primary Outcome: Change From Baseline at Day 14 for COAGULATION: Prothrombin Time and Activated Partial Thromboplastin Time
Description: Blood samples for the assessment of Prothrombin Time and Activated Partial Thromboplastin Time were collected upon participants admission to the unit.
Time Frame: Baseline and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
sec
  Baseline (Prothrombin Time ) | 11.17 (1.871) | 11.05 (1.679) | 11.91 (1.871) | 11.51 (1.757) | 11.47 (1.589)
  Day 14 Change from Baseline (Prothrombin Time) | -0.15 (0.507) | -0.32 (0.351) | 0.12 (0.503) | 0.11 (0.291) | 0.55 (2.363)
  Baseline(Activated Partial Thromboplastin Time) | 26.91 (2.435) | 27.09 (2.495) | 28.14 (2.483) | 27.50 (2.872) | 27.55 (3.009)
  Day 14 Change from Baseline (Activated Partial Thromboplastin Time): number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 Change from Baseline (Activated Partial Thromboplastin Time) | -0.82 (1.350) | -1.80 (1.489) | -0.81 (1.478) | -0.87 (1.396) | 0.58 (3.196)

41. Primary Outcome: Heart Rate (HR) - Change From Baseline (Day -1) at Day 14
Description: Heart rate was measured as part of the 12-lead electrocardiogram. Resting ECG recordings were made.Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14.
Time Frame: Baseline (day -1) and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
beats/min
  Day -1(Predose) | 65.7 (9.50) | 61.6 (6.43) | 65.3 (8.43) | 64.5 (5.85) | 65.0 (7.16)
  Day -1 (0.5 hour) | 68.5 (9.54) | 64.5 (8.76) | 66.7 (10.56) | 66.1 (9.13) | 68.7 (9.94)
  Day -1 (1 hour) | 69.8 (9.27) | 66.8 (9.58) | 66.2 (9.31) | 67.6 (5.69) | 67.2 (7.77)
  Day -1 (1.5 hour) | 68.9 (9.26) | 67.3 (7.24) | 66.5 (9.09) | 67.3 (5.38) | 67.5 (7.37)
  Day -1 (2 hour) | 70.2 (10.95) | 67.3 (7.81) | 65.9 (9.96) | 65.2 (4.38) | 66.3 (8.36)
  Day -1 (2.5 hour) | 68.7 (9.02) | 69.4 (8.86) | 64.6 (10.11) | 65.1 (4.19) | 68.2 (10.32)
  Day -1 (3 hour) | 69.4 (9.06) | 64.3 (4.91) | 65.6 (7.89) | 67.9 (5.79) | 68.8 (7.51)
  Day -1 (4 hour) | 68.0 (10.50) | 62.8 (6.70) | 64.3 (6.20) | 63.9 (5.54) | 67.5 (8.40)
  Day -1 (8 hour) | 72.9 (10.38) | 64.4 (5.95) | 70.2 (10.68) | 66.9 (7.17) | 70.2 (8.14)
  Day -1 (12 hour) | 77.0 (9.63) | 68.7 (8.96) | 73.6 (7.43) | 70.7 (7.81) | 71.6 (8.69)
  Day 14 (Pre dose) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (Pre dose) Change from Baseline | -0.4 (6.87) | -0.3 (4.08) | 0.8 (6.14) | -2.1 (6.96) | -3.8 (8.85)
  Day 14 (0.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (0.5 hour) Change from Baseline | -2.6 (7.58) | -5.1 (8.48) | -0.9 (10.10) | -4.3 (10.24) | -9.6 (10.13)
  Day 14 (1 hour) Change from Baseline | -5.0 (8.66) | -6.7 (9.65) | -0.6 (9.18) | -7.9 (8.35) | -7.7 (6.92)
  Day 14 (1.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1.5 hour) Change from Baseline | -5.5 (8.13) | -7.4 (7.24) | -1.5 (7.10) | -7.9 (8.07) | -7.6 (8.08)
  Day 14 (2 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2 hour) Change from Baseline | -6.5 (10.98) | -7.9 (7.98) | -2.4 (8.54) | -4.2 (7.90) | -7.0 (6.94)
  Day 14 (2.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2.5 hour) Change from Baseline | -4.2 (7.16) | -10.5 (8.60) | -0.3 (7.05) | -4.2 (4.95) | -7.8 (10.48)
  Day 14 (3 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (3 hour) Change from Baseline | -4.9 (9.94) | -4.6 (5.05) | -0.4 (8.45) | -7.5 (7.74) | -5.7 (9.94)
  Day 14 (4 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 13 | 15 | 13
  Day 14 (4 hour) Change from Baseline | -4.3 (8.57) | -2.9 (4.83) | 0.2 (8.86) | -2.0 (7.36) | -5.8 (7.62)
  Day 14 (8 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (8 hour) Change from Baseline | -2.2 (6.22) | 0.5 (5.15) | 6.8 (8.99) | 1.0 (6.47) | -2.3 (9.40)
  Day 14 (12 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (12 hour) Change from Baseline | -0.9 (5.70) | 0.7 (5.74) | 2.3 (8.26) | 0.0 (5.49) | -3.2 (9.57)

42. Primary Outcome: Mean PR Interval - Change From Baseline (Day -1) at Day 14
Description: PR Interval was measured as part of the 12-lead electrocardiogram. Resting ECG recordings were made. Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14.
Time Frame: Baseline (day -1) and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
msec
  Day -1 (Predose): number analyzed (Participants) | 18 | 13 | 15 | 15 | 13
  Day -1 (Predose) | 165.3 (22.20) | 152.6 (14.30) | 165.3 (26.10) | 166.6 (26.74) | 162.6 (20.52)
  Day -1 (0.5 hour) | 163.3 (24.69) | 155.3 (20.19) | 167.1 (26.74) | 162.1 (22.13) | 162.4 (20.59)
  Day -1 (1 hour) | 166.3 (23.76) | 155.7 (20.43) | 166.6 (25.79) | 166.5 (24.32) | 162.1 (19.82)
  Day -1 (1.5 hour): number analyzed (Participants) | 17 | 15 | 15 | 15 | 13
  Day -1 (1.5 hour) | 167.6 (22.91) | 158.9 (17.73) | 165.9 (21.47) | 164.9 (26.07) | 162.4 (17.60)
  Day -1 (2 hour) | 166.9 (25.01) | 156.0 (18.95) | 167.1 (22.27) | 164.9 (25.23) | 162.9 (21.16)
  Day -1 (2.5 hour): number analyzed (Participants) | 18 | 14 | 15 | 15 | 13
  Day -1 (2.5 hour) | 168.7 (26.32) | 155.3 (18.32) | 165.8 (26.24) | 165.2 (26.51) | 160.4 (21.99)
  Day -1 (3 hour) | 168.0 (25.66) | 153.7 (17.61) | 170.1 (31.39) | 161.8 (23.66) | 160.1 (20.10)
  Day -1 (4 hour) | 165.6 (24.06) | 155.4 (17.27) | 165.1 (20.73) | 163.6 (26.48) | 161.6 (16.78)
  Day -1 (8 hour) | 162.1 (23.67) | 152.5 (17.45) | 161.7 (22.93) | 163.5 (25.00) | 156.4 (16.60)
  Day -1 (12 hour) | 165.7 (26.90) | 157.7 (17.41) | 158.5 (19.56) | 159.0 (21.78) | 156.5 (17.71)
  Day 14 (Pre dose) Change from Baseline: number analyzed (Participants) | 18 | 13 | 14 | 15 | 13
  Day 14 (Pre dose) Change from Baseline | 5.6 (12.32) | 1.7 (6.41) | -1.8 (10.85) | -0.3 (9.42) | 0.9 (12.78)
  Day 14 (0.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (0.5 hour) Change from Baseline | 8.5 (20.00) | 0.4 (6.90) | 0.9 (14.64) | 4.6 (12.49) | -0.8 (13.90)
  Day 14 (1 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1 hour) Change from Baseline | 5.6 (15.88) | 2.8 (9.03) | -1.0 (14.15) | 2.7 (19.24) | 1.7 (13.74)
  Day 14 (1.5 hour) Change from Baseline: number analyzed (Participants) | 17 | 15 | 14 | 15 | 13
  Day 14 (1.5 hour) Change from Baseline | -1.0 (12.86) | -2.8 (9.59) | 3.9 (17.63) | -0.5 (11.47) | 1.8 (17.08)
  Day 14 (2 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2 hour) Change from Baseline | 4.1 (12.56) | 0.6 (8.85) | -0.9 (17.72) | 0.9 (11.82) | 4.2 (14.32)
  Day 14 (2.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2.5 hour) Change from Baseline | 2.2 (9.34) | 2.6 (13.33) | 0.0 (11.96) | 1.8 (12.11) | 8.3 (15.96)
  Day 14 (3 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (3 hour) Change from Baseline | 3.8 (11.09) | 5.3 (11.40) | -3.1 (10.83) | 4.5 (15.01) | 4.9 (14.78)
  Day 14 (4 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 13 | 13 | 13
  Day 14 (4 hour) Change from Baseline | 5.7 (15.13) | 1.4 (6.48) | 5.2 (20.77) | 1.8 (14.49) | 2.2 (9.05)
  Day 14 (8 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (8 hour) Change from Baseline | 1.4 (8.66) | 2.9 (5.95) | 0.1 (15.03) | -3.9 (12.21) | 5.2 (6.54)
  Day 14 (12 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (12 hour) Change from Baseline | -0.4 (8.83) | -3.6 (9.17) | -0.1 (11.07) | 2.0 (9.33) | 0.9 (10.80)

43. Primary Outcome: Mean QRS Duration - Change From Baseline (Day -1) at Day 14
Description: QRS Duration was measured as part of the 12-lead electrocardiogram. Resting ECG recordings were made. Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14.
Time Frame: Baseline (day -1) and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
msec
  Day -1(Predose) | 88.8 (10.82) | 93.6 (8.11) | 84.7 (6.39) | 89.2 (10.99) | 89.5 (11.76)
  Day -1 (0.5 hour | 88.7 (10.44) | 94.5 (7.94) | 87.4 (8.44) | 88.5 (10.86) | 88.9 (10.73)
  Day -1 (1 hour) | 88.7 (10.22) | 93.3 (7.17) | 85.2 (7.94) | 90.3 (9.91) | 91.2 (13.04)
  Day -1 (1.5 hour) | 89.4 (11.77) | 91.7 (8.52) | 85.0 (7.98) | 89.5 (10.20) | 92.2 (11.59)
  Day -1 (2 hour) | 86.4 (11.08) | 90.5 (7.98) | 84.0 (5.83) | 89.5 (11.15) | 89.0 (10.04)
  Day -1 (2.5 hour) | 87.6 (12.27) | 91.5 (8.94) | 84.4 (8.22) | 89.0 (10.27) | 87.8 (10.80)
  Day -1 (3 hour) | 86.4 (10.10) | 92.7 (6.94) | 85.7 (9.32) | 88.6 (10.10) | 87.9 (11.06)
  Day -1 (4 hour) | 86.2 (11.68) | 92.3 (8.26) | 85.1 (9.68) | 87.7 (11.04) | 88.7 (11.53)
  Day -1 (8 hour) | 85.4 (11.26) | 90.9 (9.16) | 81.1 (4.41) | 85.4 (11.79) | 85.3 (11.46)
  Day -1 (12 hour) | 86.6 (10.53) | 92.0 (7.93) | 85.5 (9.13) | 86.3 (10.55) | 88.1 (13.08)
  Day 14 (Pre dose) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (Pre dose) Change from Baseline | -0.7 (3.63) | 0.3 (3.89) | -0.8 (4.56) | -0.1 (6.71) | 3.1 (7.80)
  Day 14 (0.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (0.5 hour) Change from Baseline | 1.0 (7.64) | -1.2 (5.87) | -3.1 (5.37) | 0.4 (6.53) | 2.8 (5.06)
  Day 14 (1 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1 hour) Change from Baseline | 0.7 (6.66) | 0.0 (3.57) | -1.6 (7.46) | -0.1 (8.88) | -2.5 (10.73)
  Day 14 (1.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1.5 hour) Change from Baseline | -0.8 (6.00) | 1.5 (6.83) | -2.0 (6.26) | 3.4 (6.74) | -1.8 (8.62)
  Day 14 (2 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2 hour) Change from Baseline | 1.7 (8.08) | 3.2 (5.87) | -0.8 (5.25) | 1.9 (8.34) | 1.0 (8.08)
  Day 14 (2.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2.5 hour) Change from Baseline | 1.7 (7.13) | 0.9 (4.96) | 0.4 (7.02) | 1.2 (5.61) | 3.4 (7.39)
  Day 14 (3 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (3 hour) Change from Baseline | 2.2 (5.41) | 0.5 (4.87) | -1.5 (6.56) | -1.5 (7.06) | 2.6 (8.90)
  Day 14 (4 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 13 | 15 | 13
  Day 14 (4 hour) Change from Baseline | 1.9 (6.27) | 0.5 (4.61) | -2.5 (6.44) | 14.8 (49.01) | 1.7 (7.80)
  Day 14 (8 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (8 hour) Change from Baseline | -0.3 (3.82) | 1.5 (4.63) | 0.4 (3.41) | 0.9 (6.26) | 2.5 (6.05)
  Day 14 (12 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (12 hour) Change from Baseline | -1.7 (6.91) | 0.3 (2.85) | -3.3 (9.28) | -0.5 (5.49) | -0.8 (7.69)

44. Primary Outcome: Mean QT Interval - Change From Baseline (Day -1) at Day 14
Description: QT Interval was measured as part of the 12-lead electrocardiogram. Resting ECG recordings were made. Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14.
Time Frame: Baseline (day -1) and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
msec
  Day -1 (Predose) | 421.8 (31.07) | 426.4 (23.73) | 412.6 (29.12) | 421.8 (22.12) | 411.3 (16.01)
  Day -1 (0.5 hour | 412.4 (27.58) | 422.0 (24.00) | 410.1 (29.29) | 417.7 (22.13) | 405.6 (22.19)
  Day -1 (1 hour) | 412.6 (22.81) | 414.6 (21.41) | 415.6 (29.17) | 414.8 (21.32) | 406.5 (21.20)
  Day -1 (1.5 hour) | 413.7 (23.60) | 408.4 (19.91) | 408.0 (23.71) | 414.9 (21.19) | 412.3 (22.31)
  Day -1 (2 hour) | 407.4 (25.64) | 405.8 (19.18) | 410.7 (33.40) | 413.4 (20.20) | 412.7 (22.32)
  Day -1 (2.5 hour) | 411.3 (27.10) | 403.4 (27.70) | 410.9 (32.10) | 418.9 (32.10) | 412.4 (26.30)
  Day -1 (3 hour) | 407.8 (25.47) | 411.9 (22.80) | 409.9 (24.92) | 410.7 (23.04) | 401.2 (23.18)
  Day -1 (4 hour) | 408.3 (32.47) | 414.9 (20.19) | 411.2 (21.83) | 418.1 (19.01) | 407.8 (16.98)
  Day -1 (8 hour) | 398.9 (29.10) | 410.3 (19.54) | 396.3 (26.84) | 405.7 (22.57) | 398.5 (27.65)
  Day -1 (12 hour) | 389.2 (28.40) | 407.1 (22.55) | 395.5 (22.33) | 402.2 (26.39) | 394.4 (28.85)
  Day 14 (Pre dose) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (Pre dose) Change from Baseline | -6.8 (17.03) | 0.2 (15.11) | -9.6 (20.16) | -2.1 (24.54) | 5.5 (21.03)
  Day 14 (0.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (0.5 hour) Change from Baseline | 2.3 (17.73) | 8.7 (13.13) | -2.4 (23.90) | 10.2 (25.32) | 20.8 (24.94)
  Day 14 (1 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1 hour) Change from Baseline | 6.9 (18.73) | 17.8 (15.93) | -7.9 (28.71) | 16.3 (20.43) | 17.8 (22.08)
  Day 14 (1.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1.5 hour) Change from Baseline | 11.7 (22.95) | 24.5 (14.95) | -0.5 (19.09) | 15.7 (21.82) | 17.5 (21.80)
  Day 14 (2 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2 hour) Change from Baseline | 14.2 (25.19) | 25.5 (18.13) | 3.6 (25.04) | 16.3 (20.76) | 16.2 (16.67)
  Day 14 (2.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2.5 hour) Change from Baseline | 9.5 (25.18) | 28.3 (22.66) | 1.4 (24.51) | 12.9 (21.11) | 14.0 (23.04)
  Day 14 (3 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (3 hour) Change from Baseline | 14.2 (28.90) | 17.4 (15.42) | 1.9 (18.66) | 18.3 (23.65) | 17.8 (28.64)
  Day 14 (4 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 13 | 15 | 13
  Day 14 (4 hour) Change from Baseline | 12.6 (22.90) | 13.5 (15.04) | -2.8 (23.91) | 5.5 (23.97) | 18.3 (22.05)
  Day 14 (8 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (8 hour) Change from Baseline | 2.4 (14.71) | -1.9 (12.65) | -14.2 (18.23) | -3.7 (20.76) | 6.6 (27.45)
  Day 14 (12 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (12 hour) Change from Baseline | 3.0 (17.62) | -0.8 (13.58) | -12.9 (18.71) | -1.8 (16.37) | 7.8 (24.27)

45. Primary Outcome: Mean QTcF Interval (Fridericia's Correction Formula, QTcF) - Change From Baseline (Day -1) at Day 14
Description: Fridericia-corrected QTcF interval was evaluated as part of the 12-lead electrocardiogram. Resting ECG recordings were made. Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14.
Time Frame: Baseline (day -1) and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
msec
  Day -1(Predose) | 432.7 (18.75) | 429.0 (16.87) | 422.3 (14.41) | 431.1 (17.28) | 421.8 (20.02)
  Day -1 (0.5 hour) | 429.2 (16.14) | 430.9 (18.81) | 422.3 (14.40) | 430.1 (16.21) | 422.6 (15.35)
  Day -1 (1 hour) | 432.2 (14.68) | 428.3 (14.85) | 427.3 (16.15) | 430.9 (16.46) | 420.8 (13.55)
  Day -1 (1.5 hour) | 431.7 (18.47) | 423.4 (17.60) | 420.6 (14.81) | 430.5 (15.73) | 427.6 (15.24)
  Day -1 (2 hour) | 427.2 (17.33) | 420.5 (13.47) | 420.9 (15.57) | 424.5 (16.55) | 425.2 (15.08)
  Day -1 (2.5 hour) | 428.7 (19.29) | 422.1 (21.46) | 418.3 (17.41) | 429.9 (18.39) | 428.3 (17.29)
  Day -1 (3 hour) | 426.7 (16.64) | 420.3 (18.14) | 419.9 (15.56) | 427.0 (15.46) | 419.0 (17.83)
  Day -1 (4 hour) | 423.4 (19.52) | 420.3 (18.14) | 419.9 (14.74) | 426.2 (13.33) | 423.2 (19.46)
  Day -1 (8 hour) | 423.8 (16.12) | 419.3 (15.99) | 415.5 (17.53) | 419.7 (16.65) | 418.8 (25.31)
  Day -1 (12 hour) | 421.2 (16.25) | 424.2 (13.91) | 422.1 (11.25) | 423.7 (20.16) | 416.8 (20.10)
  Day 14 (Pre dose) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (Pre dose) Change from Baseline | -6.6 (11.74) | 0.3 (12.75) | -7.9 (13.31) | -6.6 (22.83) | -3.8 (13.46)
  Day 14 (0.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (0.5 hour) Change from Baseline | -3.0 (14.97) | -2.9 (9.31) | -4.4 (10.52) | 1.1 (14.51) | 0.4 (12.92)
  Day 14 (1 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1 hour) Change from Baseline | -2.6 (11.94) | 2.7 (11.08) | -8.4 (12.88) | -1.2 (18.18) | 1.6 (15.34)
  Day 14 (1.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1.5 hour) Change from Baseline | 0.1 (13.97) | 8.3 (15.45) | -3.8 (9.02) | -2.1 (15.16) | 0.6 (15.77)
  Day 14 (2 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2 hour) Change from Baseline | 1.3 (17.40) | 8.7 (11.48) | -0.4 (15.25) | 6.7 (10.09) | 0.8 (12.58)
  Day 14 (2.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2.5 hour) Change from Baseline | 1.1 (20.94) | 5.9 (18.24) | 2.3 (13.84) | 3.8 (16.62) | -2.3 (12.11)
  Day 14 (3 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (3 hour) Change from Baseline | 3.6 (13.91) | 7.0 (17.29) | 0.3 (7.71) | 2.2 (12.14) | 5.5 (15.08)
  Day 14 (4 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 13 | 15 | 13
  Day 14 (4 hour) Change from Baseline | 4.6 (11.77) | 7.1 (14.96) | -3.8 (11.34) | 0.1 (15.55) | 6.2 (22.76)
  Day 14 (8 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (8 hour) Change from Baseline | -2.0 (9.55) | -1.1 (10.67) | -1.3 (13.74) | -1.8 (14.03) | 2.0 (22.20)
  Day 14 (12 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (12 hour) Change from Baseline | 1.2 (14.43) | 1.3 (10.33) | -9.4 (13.78) | -1.3 (17.43) | 2.8 (17.21)

46. Primary Outcome: Mean QTcB Interval (Bazett's Correction Formula, QTcB) - Change From Baseline (Day -1) at Day 14
Description: Bazett-corrected QTcB interval was evaluated as part of the 12-lead electrocardiogram. Resting ECG recordings were made. Holter monitors were fitted to participants upon admission in clinic on Day -1 and Day 14.
Time Frame: Baseline (day -1) and day 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
msec
  Day -1 (Predose) | 438.6 (18.07) | 430.7 (18.10) | 427.6 (13.14) | 436.1 (17.61) | 417.3 (25.91)
  Day -1 (0.5 hour) | 438.1 (16.29) | 435.6 (21.78) | 429.1 (19.47) | 436.5 (20.61) | 431.8 (20.32)
  Day -1 (1 hour) | 442.8 (17.55) | 435.3 (18.84) | 433.7 (18.90) | 439.4 (16.23) | 428.8 (15.65)
  Day -1 (1.5 hour) | 441.3 (22.48) | 431.3 (20.62) | 427.4 (18.56) | 438.5 (15.28) | 436.0 (16.65)
  Day -1 (2 hour) | 437.8 (21.87) | 428.3 (16.51) | 426.6 (17.12) | 430.3 (16.49) | 432.1 (18.48)
  Day -1 (2.5 hour) | 438.1 (21.09) | 432.1 (22.47) | 422.7 (19.67) | 435.9 (18.04) | 436.9 (21.27)
  Day -1 (3 hour) | 436.6 (18.42) | 425.7 (22.43) | 426.7 (16.74) | 435.5 (13.93) | 428.4 (19.40)
  Day -1 (4 hour) | 431.6 (18.31) | 423.4 (21.21) | 424.6 (15.43) | 430.3 (14.06) | 431.2 (26.00)
  Day -1 (8 hour) | 437.0 (14.34) | 424.2 (17.81) | 425.9 (21.39) | 427.1 (18.11) | 429.5 (27.28)
  Day -1 (12 hour) | 438.3 (13.91) | 433.4 (16.01) | 436.4 (9.44) | 434.9 (20.98) | 428.8 (17.99)
  Day 14 (Pre dose) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (Pre dose) Change from Baseline | -6.7 (14.73) | -0.3 (13.93) | -6.9 (14.02) | -8.9 (25.90) | -8.5 (17.83)
  Day 14 (0.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (0.5 hour) Change from Baseline | -5.9 (19.59) | -8.9 (17.34) | -5.5 (13.67) | -3.4 (19.47) | -10.3 (17.32)
  Day 14 (1 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1 hour) Change from Baseline | -8.0 (16.86) | -4.6 (19.55) | -8.9 (13.33) | -10.3 (23.07) | -7.5 (16.25)
  Day 14 (1.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (1.5 hour) Change from Baseline | -6.1 (16.42) | 0.0 (21.00) | -5.5 (10.36) | -11.1 (18.95) | -8.5 (19.32)
  Day 14 (2 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2 hour) Change from Baseline | -5.7 (24.18) | -0.1 (15.10) | -2.9 (19.35) | 1.9 (13.13) | -7.5 (16.37)
  Day 14 (2.5 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (2.5 hour) Change from Baseline | -3.4 (23.12) | -5.7 (22.17) | 2.2 (15.76) | -1.4 (17.37) | -10.8 (16.97)
  Day 14 (3 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (3 hour) Change from Baseline | -1.6 (13.90) | 1.9 (20.81) | -0.4 (11.01) | -6.3 (12.49) | -0.7 (14.57)
  Day 14 (4 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 13 | 15 | 13
  Day 14 (4 hour) Change from Baseline | 0.4 (13.21) | 3.3 (17.73) | -4.2 (12.68) | -2.2 (16.13) | -0.1 (27.06)
  Day 14 (8 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (8 hour) Change from Baseline | -4.4 (12.46) | -0.8 (13.48) | 5.5 (19.09) | -0.9 (14.17) | -0.2 (24.65)
  Day 14 (12 hour) Change from Baseline: number analyzed (Participants) | 18 | 15 | 14 | 15 | 13
  Day 14 (12 hour) Change from Baseline | 0.3 (15.11) | 2.1 (13.19) | -7.5 (16.64) | -1.2 (20.57) | -0.2 (18.66)

47. Primary Outcome: Nature and Severity of Adverse Events (AEs) up to Day 21
Description: An AE was defined as any untoward medical occurrence in a subject or clinical trial subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product.
  Serious Adverse Event (SAE) is an adverse event that at any dose: Results in death, Is life-threatening (i.e. the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it was more severe), Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, Is considered to be an important medical event.
Time Frame: On or after first drug administration up to end of study (Day 21).
Measure: Number; unit: Participants
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Participants
  Any TEAE | 13 | 7 | 11 | 10 | 11
  Any Mild TEAE | 12 | 7 | 10 | 10 | 11
  Any Moderate TEAE | 1 | 1 | 1 | 1 | 1
  Any Severe TEAE | 0 | 0 | 0 | 0 | 0
  Any serious TEAE | 9 | 7 | 7 | 5 | 11
  Any Causally Related TEAE | 9 | 7 | 7 | 5 | 11
  Any Causally Related Serious TEAE | 11 | 0 | 0 | 0 | 0
  Any Life Threatening Serious TEAE | 0 | 0 | 0 | 0 | 0
  Any TEAE of Dehydration | 0 | 0 | 0 | 0 | 0
  Any Death | 0 | 0 | 0 | 0 | 0

48. Primary Outcome: Withdrawals Due to AEs up to Day 21
Description: as for outcome 47
Time Frame: On or after first drug administration up to end of study (Day 21)
Measure: Number; unit: Participants
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Participants
  Any TEAE Leading to Discontinuation of Study Drug | 0 | 0 | 0 | 0 | 0
  Any TEAE Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Change in Frequency of Hot Flushes From Baseline (Day -1) at Days 7, 14 as Assessed by Skin Conductance
Description: Sternal skin conductance monitors (the Bahr MonitorTM) and the associated algorithm software were supplied by Simplex Scientific LLC (Middleton, USA).
  Participants were instructed to push a button on the skin conductance monitor when they sensed a hot flush when fitted with the monitor and then provide details of the hot flush in the continuous hot flush diary. Sternal skin conductance monitors were fitted on Day -1 (24 hours±1 hour prior to the planned study drug administration on Day 1) and remained in place until after the Day 7 24-hour assessments were completed (on Day 8). Refitted around 30 minutes prior to study drug administration on Day 14 and remained in place until after the 24-hour assessments were completed on Day 15.
Time Frame: Baseline (day -1) and days 7, 14
Population: Participants with available data reported.
Measure: Mean (Standard Deviation); unit: Hot flushes
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Hot flushes
  Baseline ( Day -1): number analyzed (Participants) | 17 | 12 | 14 | 15 | 12
  Baseline ( Day -1) | 5.486 (7.148) | 8.680 (4.720) | 7.787 (6.153) | 3.200 (4.945) | 5.583 (7.242)
  Change from Day -1 to Day 7: number analyzed (Participants) | 15 | 5 | 14 | 12 | 7
  Change from Day -1 to Day 7 | -0.857 (6.794) | -3.986 (6.487) | -3.679 (4.670) | -2.197 (4.6090) | 0.000 (6.2450)
  Change from Day -1 to day 14: number analyzed (Participants) | 14 | 12 | 13 | 10 | 11
  Change from Day -1 to day 14 | -0.139 (8.0619) | -2.642 (6.0682) | -2.913 (6.4202) | 0.600 (4.9261) | -2.908 (7.1204)

50. Secondary Outcome: Change From Baseline (Week -1) at Weeks 1, 2 in Frequency of Moderate to Severe Hot Flushes as Measured by Twice Daily Paper Diary Throughout Study
Description: Hot flush frequency and hot flush severity were obtained using the Hot Flush paper Diary. Subjects documented the number of individual hot flushes experienced and rated the severity of each on a scale of 1 to 3 (mild = 1, moderate = 2, severe = 3). The diaries were completed based on recall twice daily, in the morning and evening.
Time Frame: Baseline (week -1) and Week 1 ,Week 2
Measure: Mean (Standard Deviation); unit: Hot flushes
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Hot flushes
  Baseline (Week -1) | 10.44 (3.866) | 12.70 (3.385) | 12.04 (3.606) | 10.22 (2.976) | 9.90 (2.107)
  Change from Week -1 to Week 1 | -2.53 (3.645) | -1.91 (4.610) | -5.35 (5.153) | -6.36 (3.818) | -4.49 (2.801)
  Change from Week -1 to Week 2 | -3.87 (4.179) | -3.07 (5.647) | -7.09 (4.915) | -8.62 (3.749) | -6.54 (3.453)

51. Secondary Outcome: Change From Baseline (Week -1) at Weeks 1, 2 in Average Daily Severity of Hot Flushes as Measured by Twice Daily Paper Diary
Description: Participants documented the number of individual hot flushes experienced and rated the severity of each on a scale of 1 to 3 (mild = 1, moderate = 2, severe = 3). The diaries were completed based on recall twice daily, in the morning and evening.
Time Frame: Baseline (week -1) and weeks 1, Week 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Scores on a scale
  Week -1 | 2.32 (0.304) | 2.31 (0.319) | 2.20 (0.267) | 2.16 (0.379) | 2.19 (0.304)
  Change from Week -1 to Week 1 | -0.30 (0.358) | -0.21 (0.276) | -0.23 (0.318) | -0.51 (0.542) | -0.34 (0.533)
  Change from Week -1 to Week 2 | -0.34 (0.383) | -0.23 (0.242) | -0.36 (0.359) | -0.88 (0.656) | -0.42 (0.757)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.4641, Linear mixed-effects model; LS means difference = 0.09, 90% CI 2-sided [-0.12 to 0.30], Standard Error of Mean 0.127 — Change from Week -1 to Week 1
Statistical Analysis 2: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.9894, LS means difference; Linear mixed-effects model = 0.00, 90% CI 2-sided [-0.21 to 0.21], Standard Error of Mean 0.128 — Change from Week -1 to Week 1
Statistical Analysis 3: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0199, Linear mixed-effects model; LS means difference = -0.31, 90% CI 2-sided [-0.52 to -0.09], Standard Error of Mean 0.129 — Change from Week -1 to Week 1
Statistical Analysis 4: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.3907, Linear mixed-effects model; LS means difference = -0.12, 90% CI 2-sided [-0.34 to 0.11], Standard Error of Mean 0.133 — Change from Week -1 to Week 1
Statistical Analysis 5: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.5393, Linear mixed-effects model; LS means difference = 0.10, 90% CI 2-sided [-0.17 to 0.38], Standard Error of Mean 0.166 — Change from Week -1 to Week 2
Statistical Analysis 6: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.7931, Linear mixed-effects model; LS means difference = -0.04, 90% CI 2-sided [-0.33 to 0.24], Standard Error of Mean 0.169 — Change from Week -1 to Week 2
Statistical Analysis 7: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0004, Linear mixed-effects model; LS means difference = -0.63, 90% CI 2-sided [-0.92 to -0.35], Standard Error of Mean 0.169 — Change from Week -1 to Week 2
Statistical Analysis 8: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.3739, Linear mixed-effects model; LS means difference = -0.16, 90% CI 2-sided [-0.45 to 0.13], Standard Error of Mean 0.175 — Change from Week -1 to Week 2

52. Secondary Outcome: Change From Baseline (Week -1) at Weeks 1, 2 in Average Daily Hot Flushes Severity Score as Measured by Twice Daily Paper Diary.
Description: The hot flushes severity score was a composite of the frequency and severity of hot flushes, and was calculated as follows: number of mild hot flushes recorded on Day Y + number of moderate hot flushes recorded on Day Y × 2 + number of severe hot flushes recorded on Day Y × 3. Higher scores mean more severe hot flushes.
Time Frame: Baseline (week -1) and week 1 , 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Scores on a scale
  Week -1 | 28.06 (11.631) | 33.74 (8.875) | 32.52 (11.203) | 27.87 (7.720) | 26.75 (5.416)
  Change from Week -1 to Week 1 | -6.99 (9.673) | -5.56 (10.907) | -14.48 (14.275) | -17.03 (9.996) | -12.23 (7.284)
  Change from Week -1 to Week 2 | -10.67 (10.542) | -8.02 (13.031) | -19.19 (14.211) | -22.82 (9.505) | -17.55 (8.953)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0900, Linear mixed-effects model; LS means difference = 5.29, 90% CI 2-sided [0.16 to 10.42], Standard Error of Mean 3.077 — Change from Week -1 to Week 1
Statistical Analysis 2: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.1487, Linear mixed-effects model; LS means difference = -4.46, 90% CI 2-sided [-9.55 to 0.63], Standard Error of Mean 3.053 — Change from Week -1 to Week 1
Statistical Analysis 3: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0012, Linear mixed-effects model; LS means difference = -10.18, 90% CI 2-sided [-15.20 to -5.15], Standard Error of Mean 3.015 — Change from Week -1 to Week 1
Statistical Analysis 4: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0548, Linear mixed-effects model; LS means difference = -6.14, 90% CI 2-sided [-11.37 to -0.90], Standard Error of Mean 3.142 — Change from Week -1 to Week 1
Statistical Analysis 5: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0522, Linear mixed-effects model; LS means difference = 6.59, 90% CI 2-sided [1.03 to 12.15], Standard Error of Mean 3.337 — Change from Week -1 to Week 2
Statistical Analysis 6: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.1326, Linear mixed-effects model; LS means difference = -5.07, 90% CI 2-sided [-10.61 to 0.48], Standard Error of Mean 3.329 — Change from Week -1 to Week 2
Statistical Analysis 7: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0004, Linear mixed-effects model; LS means difference = -12.28, 90% CI 2-sided [-17.73 to -6.83], Standard Error of Mean 3.270 — Change from Week -1 to Week 2
Statistical Analysis 8: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0253, Linear mixed-effects model; LS means difference = -7.79, 90% CI 2-sided [-13.47 to -2.11], Standard Error of Mean 3.408 — Change from Week -1 to Week 2

53. Secondary Outcome: Change in Frequency From Baseline (Day -1), at Days 7, 14 of Hot Flushes as Measured by Continuous Day Time Diary.
Description: Subjects recorded each hot flush and its severity on a scale of 1 to 3 (mild = 1, moderate = 2, severe = 3) in the hot flush paper diary as they occurred during the day and night.
Time Frame: Baseline(day -1) and Day 7, 14
Population: Participants with available data reported.
Measure: Least Squares Mean (90% Confidence Interval); unit: Hot flushes
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Hot flushes
  Day 7 Change from Day -1 | -2.8 [-4.5 to -1.0] | -1.4 [-3.4 to 0.6] | -5.1 [-7.0 to -3.2] | -8.3 [-10.2 to -6.4] | -5.8 [-7.9 to -3.8]
  Day 14 Change from Day -1 | -3.6 [-4.9 to -2.2] | -2.3 [-3.8 to -0.8] | -6.0 [-7.5 to -4.5] | -8.6 [-10.0 to -7.1] | -7.0 [-8.6 to -5.4]
Statistical Analysis 1: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.3796, Linear mixed-effects model; LS means difference = 1.4, 90% CI 2-sided [-1.2 to 4.0], Standard Error of Mean 1.58 — Day 7 Change from Day -1
Statistical Analysis 2: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.1413, Linear mixed-effects model; LS means difference = -2.3, 90% CI 2-sided [-4.9 to 0.3], Standard Error of Mean 1.55 — Day 7 Change from Day -1
Statistical Analysis 3: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0007, Linear mixed-effects model; LS means difference = -5.5, 90% CI 2-sided [-8.1 to -2.9], Standard Error of Mean 1.55 — Day 7 Change from Day -1
Statistical Analysis 4: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0624, Linear mixed-effects model; LS means difference = -3.1, 90% CI 2-sided [-5.8 to -0.4], Standard Error of Mean 1.62 — Day 7 Change from Day -1
Statistical Analysis 5: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.2930, Linear mixed-effects model; LS means difference = 1.3, 90% CI 2-sided [-0.7 to 3.3], Standard Error of Mean 1.21 — Day 14 Change from Day -1
Statistical Analysis 6: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0512, Linear mixed-effects model; LS means difference = -2.4, 90% CI 2-sided [-4.4 to -0.4], Standard Error of Mean 1.21 — Day 14 Change from Day -1
Statistical Analysis 7: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p < 0.0001, Linear mixed-effects model; LS means difference = -5.0, 90% CI 2-sided [-7.0 to -3.0], Standard Error of Mean 1.20 — Day 14 Change from Day -1
Statistical Analysis 8: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0080, Linear mixed-effects model; LS means difference = -3.4, 90% CI 2-sided [-5.5 to -1.3], Standard Error of Mean 1.25 — Day 14 Change from Day -1

54. Secondary Outcome: Change From Baseline (Week -1) at Weeks 1, 2 in Night-time Awakenings (NTA) Secondary to Hot Flushes as Measured by Paper Diary
Description: The number of NTAs secondary to hot flushes was the sum of the number of moderate and severe night-time hot flushes recorded the following morning (twice-daily hot flush diary) or recorded contemporaneously on the continuous diary.
Time Frame: Baseline (week-1) and weeks 1 , 2
Measure: Mean (Standard Deviation); unit: Night-time Awakenings
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
Night-time Awakenings
  Baseline (Week -1) | 4.51 (2.282) | 5.61 (1.785) | 5.41 (2.337) | 4.74 (2.111) | 4.76 (1.443)
  Change from Week -1 to Week 1 | -0.77 (2.066) | -0.80 (2.448) | -2.52 (2.604) | -2.75 (2.335) | -2.07 (1.833)
  Change from Week -1 to Week 2 | -1.44 (2.128) | -1.12 (2.665) | -3.00 (2.751) | -3.83 (2.008) | -3.02 (2.117)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.1482, Linear mixed-effects model; LS means difference = 0.84, 90% CI 2-sided [-0.12 to 1.80], Standard Error of Mean 0.574 — Change from Week -1 to Week 1
Statistical Analysis 2: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0734, Linear mixed-effects model; LS means difference = -1.04, 90% CI 2-sided [-1.99 to -0.09], Standard Error of Mean 0.571 — Change from Week -1 to Week 1
Statistical Analysis 3: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0022, Linear mixed-effects model; LS means difference = -1.80, 90% CI 2-sided [-2.74 to -0.86], Standard Error of Mean 0.565 — Change from Week -1 to Week 1
Statistical Analysis 4: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0660, Linear mixed-effects model; LS means difference = -1.10, 90% CI 2-sided [-2.08 to -0.12], Standard Error of Mean 0.589 — Change from Week -1 to Week 1
Statistical Analysis 5: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0593, Linear mixed-effects model; LS means difference = 1.18, 90% CI 2-sided [0.15 to 2.20], Standard Error of Mean 0.613; Change from Week -1 to Week 2
Statistical Analysis 6: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other; p = 0.1354, Linear mixed-effects model; LS means difference = -0.93, 90% CI 2-sided [-1.95 to 0.10], Standard Error of Mean 0.614 — Change from Week -1 to Week 2
Statistical Analysis 7: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0005, Linear mixed-effects model; LS means difference = -2.20, 90% CI 2-sided [-3.21 to -1.20], Standard Error of Mean 0.603 — Change from Week -1 to Week 2
Statistical Analysis 8: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive Analysis; p = 0.0309, Linear mixed-effects model; LS means difference = -1.38, 90% CI 2-sided [-2.43 to -0.34], Standard Error of Mean 0.628 — Change from Week -1 to Week 2

55. Secondary Outcome: Change From Baseline (Day-1) to Day 1 and Day 7 in Luteinizing Hormone (AUC0-8)
Description: Change in Luteinizing Hormone(LH) AUC from time zero to 8 hours. Pre-dose samples for LH were taken within 30 minutes prior to dose administration.
Time Frame: baseline (day-1) to day 1 and day 7, pre-dose and post-dose (0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 5.0, 6.0, 8.0, 12.0 and 24.0 hours)
Measure: Mean (Standard Deviation); unit: h*U/L
Arm/Group | Placebo | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
Number analyzed (Participants) | 18 | 15 | 15 | 15 | 13
h*U/L
  Day -1 | 295.4 (82.64) | 295.5 (85.22) | 290.8 (85.83) | 309.5 (104.38) | 261.1 (65.53)
  Change from Day -1 to Day 1 | 14.4 (31.33) | 4.7 (35.80) | -10.0 (21.90) | -31.1 (38.28) | -24.6 (32.36)
  Change from Day -1 to Day 7 | 12.4 (57.46) | 22.9 (37.07) | 10.2 (20.49) | -12.1 (47.30) | -4.4 (33.43)
Statistical Analysis 1: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.3768, Linear mixed-effects model; LS means difference = -9.7, 90% CI 2-sided [-27.8 to 8.5], Standard Error of Mean 10.88 — Change from Day -1 to Day 1
Statistical Analysis 2: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.0248, Linear mixed-effects model; LS means difference = -25.0, 90% CI 2-sided [-43.1 to -6.8], Standard Error of Mean 10.89 — Change from Day -1 to Day 1
Statistical Analysis 3: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.0001, Linear mixed-effects model; LS means difference = -43.9, 90% CI 2-sided [-62.1 to -25.8], Standard Error of Mean 10.90 — Change from Day -1 to Day 1
Statistical Analysis 4: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.0004, Linear mixed-effects model; LS means difference = -42.9, 90% CI 2-sided [-61.9 to -23.8], Standard Error of Mean 11.43 — Change from Day -1 to Day 1
Statistical Analysis 5: Comparison: Placebo vs 50 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.4819, Linear mixed-effects model; LS means difference = 10.4, 90% CI 2-sided [-14.2 to 35.1], Standard Error of Mean 14.76 — Change from Day -1 to Day 7
Statistical Analysis 6: Comparison: Placebo vs 100 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.8694, Linear mixed-effects model; LS means difference = -2.4, 90% CI 2-sided [-27.1 to 22.2], Standard Error of Mean 14.77 — Change from Day -1 to Day 7
Statistical Analysis 7: Comparison: Placebo vs 150 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.1105, Linear mixed-effects model; LS means difference = -23.9, 90% CI 2-sided [-48.6 to 0.7], Standard Error of Mean 14.79 — Change from Day -1 to Day 7
Statistical Analysis 8: Comparison: Placebo vs 300 mg BAY3427080; Test type: Other — Descriptive analysis; p = 0.2390, Linear mixed-effects model; LS means difference = -18.4, 90% CI 2-sided [-44.2 to 7.4], Standard Error of Mean 15.50 — Change from Day -1 to Day 7

ADVERSE EVENTS:
Time Frame: Adverse events data were collected on or after first drug administration up to end of study (Day 21).
Groups:
- Placebo Comparator: Placebo to match BAY3427080 (NT-814) capsules administered orally, daily, for 14 days. Number of placebo capsules to match active dose.
Arm/Group | Placebo Comparator | 50 mg BAY3427080 | 100 mg BAY3427080 | 150 mg BAY3427080 | 300 mg BAY3427080
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/15 | 0/15 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/15 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 13/18 | 7/15 | 11/15 | 10/15 | 11/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator (N=18) | 50 mg BAY3427080 (N=15) | 100 mg BAY3427080 (N=15) | 150 mg BAY3427080 (N=15) | 300 mg BAY3427080 (N=13)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Medical device site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (1) | 6 (6)
Somnolence (Nervous system disorders) | 3 (3) | 5 (5) | 2 (2) | 5 (5) | 9 (11)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 6 (6) | 5 (5) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is required to postpone communication of results until a joint, multicenter publication of the multicenter study has occurred, or the sponsor confirms that no joint publication will be prepared, or 18 months since completion of the data analysis have passed.

The sponsor can review planned publications for up to 60 days and request reasonable amendments. The review period can be extended by up to 6 months in case a patent application is planned.

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT02865538/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT02865538/SAP_001.pdf